CLINICAL TRIAL: NCT05060783
Title: Renal Cancer Detection With Liquid Biopsy
Acronym: GaGnostic
Status: Recruiting | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: Lund University (Other); Elypta (Industry)
Responsible Party: Principal Investigator, Nessn Azawi, Associate professor, Zealand University Hospital
Other Study IDs: SJ-894
Record Dates: First submitted 2021-09-16; First posted 2021-09-29 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Renal Cancer; Oncocytoma
MeSH Terms: conditions — Kidney Neoplasms; Adenoma, Oxyphilic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Serum and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Renal Call Carcinoma: Patrients with renal cancer
  Interventions: Diagnostic Test: GaGnostic
- Oncocytoma: Patients with oncocytoma
  Interventions: Diagnostic Test: GaGnostic
- Healthy persons: Patients with CT scan shows no renal cancer
  Interventions: Diagnostic Test: GaGnostic

INTERVENTIONS:
Diagnostic Test: GaGnostic — Plasma
  Other Names: Glycosaminoglycan
Diagnostic Test: GaGnostic — Serum
  Other Names: Glycosaminoglycan
Diagnostic Test: GaGnostic — Urine
  Other Names: Glycosaminoglycan

SUMMARY:
Glycosaminoglycans (GAGs) were significantly altered in localized as well advanced RCC compared to healthy samples. In addition, GAG scores correlated with progression-free survival and overall survival (OS) in a prospective cohort of patients with metastatic ccRCC and localized RCC. However, it is still unknown whether alterations in plasma and urine GAGs are exquisitely specific to RCC or are shared by other benign lesions in the kidney, such as angiomyolipomas, oncocytomas, or PEComa.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent CT-scan with suspicion of renal tumor and the scans show no sign of renal cancer.
2. For patient with ccRCC or oncocytoma, they should have a histological verified tumor (Biopsy or surgical specimen)
3. Sign up information consent
4. Can perform protocol procedure

Exclusion Criteria:

1. Non-clear cell Renal cell carcinoma
2. RCC with pure sarcomatoid differentiation, also called sarcoma of the kidney
3. Use of heparin for concurrent disease in need of blood dilution (e.g. ongoing deep vein thrombosis or lung emboli). Note: use of of heparin for thrombus prophylaxis in conjunction with primary surgery or postoperatively ≤4 weeks will be allowed.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients referred to our department by family doctors or the primary sector with a suspicion of renal tumor by CT-scanning will be asked to participate in the study. Patients with suspected small renal tumor will be offered renal tumor biopsies as standard procedure.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
To identify the optimal GAG score | 2 years
  To identify the optimal GAG score in RCC patients
To identify the optimal GAG score | 2 years
  To identify the optimal GAG score in oncocytoma
To identify the optimal GAG score | 2 years
  To identify the optimal GAG score in healthy individuel

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: Undecided